CLINICAL TRIAL: NCT00505544
Title: The Brief Sleep Disturbance Scale: Measuring Sleep Disturbance Among Cancer Patients
Brief Title: Measuring Sleep Disturbance Among Cancer Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-0598
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Advanced Cancer
Keywords: Advanced Cancer; Questionnaire; Survey; Sleep Disturbance; Sleep Quality
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Questionnaire: Questionnaires that ask about your sleep, symptoms, and mood.
  Interventions: Behavioral: Questionnaire
- Questionnaire + Actigraphs: Questionnaires that ask about your sleep, symptoms, and mood. Wear actigraph to collect information on activity levels and sleep patterns for one week.
  Interventions: Behavioral: Questionnaire; Device: Actigraph

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires that ask about your sleep, symptoms, and mood.
  Other Names: Survey
Device: Actigraph — Wear actigraph to collect information on activity levels and sleep patterns for one week.
  Groups: Questionnaire + Actigraphs

SUMMARY:
Objectives:

Primary Objectives:

1. To establish concurrent criterion-related validity of the Brief Sleep Disturbance Scale (BSDS) by correlating the scale with the Pittsburgh Sleep Quality Index.
2. To evaluate the construct validity of the BSDS through exploratory factor analysis.
3. To examine possible predictors of sleep disturbance.
4. To evaluate the reliability of the BSDS using Cronbach's coefficient alpha and test-retest reliability.
5. To evaluate the sensitivity of the BSDS by administering it to the same group of patients (n = 60) prior to treatment with a regimen associated with sleep disturbance, during 4 weeks of treatment, and upon completion of treatment.
6. To evaluate the psychometric properties of the BSDS in a sample of community dwelling adults.

Secondary Objective:

1. To obtain pilot data from a small sample of patients who will wear an actigraph for one week.

DETAILED DESCRIPTION:
Patients Who Complete the Surveys on Multiple Time Points:

This study will teach researchers about changes in your sleep patterns that may happen during your cancer treatment. The participants will be recruited from the Melanoma Clinic.

If you agree to take part in this study, during your cancer treatment, you will be asked to complete three written questionnaires that ask about your sleep, symptoms, and mood. These questionnaires will take about 20 minutes to complete. You will be asked to complete the questionnaires before, during and after your cancer treatment during 11 of your clinic visits.

You will also be asked to fill out a sleep diary at home, in which you will be asked to record what time you go to bed, whether you get up during the night, and what time you wake up. You will be asked to fill out the diary every day, for one week. You will be asked to return it during a clinic visit or by mail, with a stamped envelope that will be provided.

During the study, the research staff will collect information from your medical chart about your cancer, cancer treatment, and laboratory tests.

This is an investigational study. Up to 570 participants will take part in this multicenter study. Up to 380 will be enrolled at MD Anderson.

Patients Who Wear Actigraphs:

This study will help researchers to understand how cancer and cancer treatments affect sleep patterns. The participants will be recruited from the M. D. Anderson outpatient clinics, including Breast, Neuro-oncology, Blood and Marrow Transplantation, Genitourinary Oncology, Gastrointestinal Oncology Gynecologic Oncology, Head and Heck, Thoracic Oncology, Leukemia, Lymphoma, Melanoma, Sarcoma, Internal Medicine, and the Ambulatory Treatment Center.

If you agree to take part in this study, you will be asked to complete eight written questionnaires that have questions about your sleep, symptoms, and mood. These questionnaires will take about 20 minutes to complete. You will be asked to fill out the questionnaires before wearing the actigraph and after one week of wearing the actigraph.

During the study, the research staff will collect information from your medical chart about the cancer, cancer treatment, and laboratory tests.

You will be asked to wear an actigraph on your wrist for one week. An actigraph is a small motion detector that is about the size and shape of a wristwatch. The actigraph will collect and store information on your activity levels and your sleep patterns. You will be asked to return the actigraph at the end of the week.

You will be asked to fill out a sleep diary at home, in which you will be asked to record what time you go to bed, whether you get up during the night, and what time you wake up. You will only be asked to do this during the week you wear the actigraph.

At the end of the "actigraph" week, you will be asked to complete a brief sleep questionnaire, which will take about 5 minutes to complete.

This is an investigational study. About 20 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient or inpatient receiving evaluation, treatment, or follow-up care at MDACC or a collaborating site.
2. Has a pathological diagnosis of cancer.
3. 18 years of age or older.
4. Able to understand English.
5. Gives informed consent to participate.
6. Community sample eligibility: Community dwelling adult who attends a meeting of a designated service organization.
7. Community sample eligibility: 18 years of age or older
8. Community sample eligibility: Gives Informed Consent to participate.
9. Community sample eligibility: Able to understand English.

Exclusion Criteria:

1. Cannot understand the intent of the study.
2. Patient feels too ill to complete the surveys.
3. Refuses to participate.
4. Community sample exclusion criterion: Unable to complete the surveys.
5. Community sample exclusion criterion: Refuses to participate.
6. Community sample exclusion criterion: Cancer diagnosis (past or present).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants with a pathological diagnosis of cancer and community dwelling adults who attend a meeting of a designated service organization.
Sampling Method: Non-Probability Sample
Enrollment: 459 (Actual)
Dates: Start 2005-08 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Brief Sleep Disturbance Scale (BSDS) | Administering to same group prior to treatment with a regimen associated with sleep disturbance, during 4 weeks of treatment, and upon completion of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xin S. Wang, MD,MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org